CLINICAL TRIAL: NCT03103386
Title: Effects of Fermented Rye Bran Products on HP Infection and Metabolic Risk Factors
Brief Title: Effects of Fermented Rye Bran Products on Helicobacter Pylori (HP) Infection and Metabolic Risk Factors
Acronym: RyeClaim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Collaborators: Swedish University of Agricultural Sciences (Other); Shanghai Zhongye Hospital (Unknown)
Responsible Party: Principal Investigator, Gengsheng He, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KEF201196
Record Dates: First submitted 2016-12-23; First posted 2017-04-06 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: H. Pylori Infections; Non-communicable Diseases
Keywords: fermented rye bran; H. pylori infections; non-communicable diseases
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fermented Rye Bran group (Experimental): Intake of food product with a patented fermented rye bran: A patented fermented rye bran ingredient for food purpose has been produced through a process where a specific Lactobacillus curvatis strain was incubated with rye bran by Kampffmayer Food Innovation GmbH, Germany. The dried fermented rye bran was incorporated into a whole grain rye crisp bread product (25% on weight basis) commercially available in Sweden and in a novel extruded whole grain rye product (20%) developed by Lantmännen.Two crisp rye bread pieces (2 x 12g) were packed into moisture and air tight portion package. Participants are advised to consume 4 pieces daily. Rye puff was packed into 2 moisture and air tight portion bags. Participants are advised to consume 2 bags daily. Total energy: 518 kcal/day.
  Interventions: Dietary Supplement: intake of food product with a patented fermented rye bran
- Refined Wheat group (Placebo Comparator): Intake of food product with common refined wheat: Corresponding crisp bread and extruded product will be produced using refined wheat flour. Two crisp bread pieces (2 x 12 g) were packed into moisture and air tight portion package. Participants are advised to consume 4 pieces daily.Wheat puff was packed into 2 moisture and air tight portion bags. Participants are advised to consume 2 bags daily.Total energy: 513 kcal/day.
  Interventions: Dietary Supplement: intake of food product with common refined wheat

INTERVENTIONS:
Dietary Supplement: intake of food product with a patented fermented rye bran — During the treatment period, participants will be provided 2 packages of puff（fermented rye bran）and 2 packages of crisp bread to be included in the daily diet. Participants are free to consume the product any time during the day to facilitate compliance.
  Arms: Fermented Rye Bran group
Dietary Supplement: intake of food product with common refined wheat — During the treatment period, participants will be provided 2 packages of puff （common refined wheat）and 2 packages of crisp bread to be included in the daily diet. Participants are free to consume the product any time during the day to facilitate compliance.
  Arms: Refined Wheat group

SUMMARY:
The investigators hypothesize that long-term fermented high-fibre rye intake may reduce the Helicobacter pylori infection through dampening inflammation and thereby leading to lower adherence of the bacteria to surfaces.The investigators further hypothesize that that inflammation could be a potential causal link between HP infection and insulin resistance, a risk factor for type 2 diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
A randomized, double-blind, 12 week parallel dietary intervention study is conducted to evaluate the effects of the two novel food products containing fermented rye bran in normal weight and overweight men and women with prevalent HP infection. A follow-up is planned at week 24. The primary endpoint is severity of HP infection indicated by a breath test. Secondary endpoints include effects on chronic inflammation, insulin resistance, blood lipids, blood cholesterol,body weight, intestinal microbial clusters et al. The food products given to the treatment group will be a novel breakfast cereal product and a crispbread product containing fermented rye bran. The control product will be corresponding products based on refined wheat.

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women are eligible.
2. Age: 20-70 years old.
3. HP: 13C-urea breath test value（DOB）above 4.
4. 50% of the participants should have BMI below or equal to 24 and 50% should have BMI above 24.
5. Willing to consume test products for 12 weeks.

Exclusion Criteria:

1. Smokers.
2. In medication (except medication for mild hypertension).
3. Having allergies or food intolerance.
4. Having chronic disease, such as type 2 diabetes, cardiovascular disease and cancer.
5. Diagnosis of peptic ulcer.
6. Pregnancy or to be pregnant.
7. Having travel plans in 4 months.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
HP infection | 6，12 and 24 weeks
  The primary endpoint is the changes of severity of HP infection indicated by a C13-ureabreath test

SECONDARY OUTCOMES:
Analyzes of chronic inflammation | Up to 10 months
  Analyzes of IL-1, IL-2, IL-6, IL-8, IL-10, inf-γ and hs-CRP with 100 µl plasma or serum
Analyzes of blood lipids | 6，12 and 24 weeks
  Analyzes of the changes of total cholesterol, HDL/LDL and TAG with 100 µl serum
Analyzes of blood glucose and insulin | 6，12 and 24 weeks
  Analyzes of the changes of glucose, insulin and HOMA-IR with 150 µl serum or plasma
Analyzes of alkylresorcinols | Up to 10 months
  Biomarkers of whole grain wheat and rye intake, 200 µl plasma or serum
Analyzes of body weight changes | 6，12 and 24 weeks
Analyzes of gut microbiota | Up to 2 years
  Analyzes of 16S rDNA by Illumina MiSeq with feces

CONTACTS AND LOCATIONS:
Overall Officials: Gengsheng He, PhD., Principal Investigator — Fudan University
Locations (1):
- Dept. Nutrition and Food Hygiene, School of Public Health,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polyzos SA, Kountouras J, Zavos C, Deretzi G. The association between Helicobacter pylori infection and insulin resistance: a systematic review. Helicobacter. 2011 Apr;16(2):79-88. doi: 10.1111/j.1523-5378.2011.00822.x. PMID 21435084
- [Background] Landberg R, Andersson SO, Zhang JX, Johansson JE, Stenman UH, Adlercreutz H, Kamal-Eldin A, Aman P, Hallmans G. Rye whole grain and bran intake compared with refined wheat decreases urinary C-peptide, plasma insulin, and prostate specific antigen in men with prostate cancer. J Nutr. 2010 Dec;140(12):2180-6. doi: 10.3945/jn.110.127688. Epub 2010 Oct 27. PMID 20980650
- [Background] McKeown NM, Troy LM, Jacques PF, Hoffmann U, O'Donnell CJ, Fox CS. Whole- and refined-grain intakes are differentially associated with abdominal visceral and subcutaneous adiposity in healthy adults: the Framingham Heart Study. Am J Clin Nutr. 2010 Nov;92(5):1165-71. doi: 10.3945/ajcn.2009.29106. Epub 2010 Sep 29. PMID 20881074
- [Derived] Xue K, Liu Y, Iversen KN, Mazidi M, Qu Z, Dong C, Jin T, Hallmans G, Aman P, Johansson A, He G, Landberg R. Impact of a Fermented High-Fiber Rye Diet on Helicobacter pylori and Cardio-Metabolic Risk Factors: A Randomized Controlled Trial Among Helicobacter pylori-Positive Chinese Adults. Front Nutr. 2021 Jan 15;7:608623. doi: 10.3389/fnut.2020.608623. eCollection 2020. PMID 33521037